CLINICAL TRIAL: NCT06778733
Title: The Effect of Clomiphene Citrate Administration in Combination with Low Dose (150 IU) of Gonadotropins Vs High Dose Gonadotropin Protocol in Poor Responders. Impact on Stimulation Characteristics and Pregnancy Outcome.
Brief Title: Effectiveness of Low Dose Gonadotropin Stimulation Protocol Vs High Dose Gonadotropin Protocol in Poor Responders
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Nikos Vlahos, Professor of Obstetrics and Gynecology, Head of the Department, Aretaieion University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARETAIEION IVF UNIT
Record Dates: First submitted 2024-10-05; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Female Infertility
Keywords: Clomiphene Citrate; IVF; Gonadotrophins; pregnancy rates; ovarian reserve; Low-dose gonadotrophins
MeSH Terms: conditions — Infertility, Female | interventions — Clomiphene; follitropin alfa

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Clomiphene Citrate (CC)/r-FSH (Active Comparator): Administration of 100mg/day Clomiphene citrate (CC) from day 3 to day 7 of the cycle (5 days) in combination with low-dose gonadotropins (150IU) according to a short stimulation GnRh antagonists protocol.
  Treatment schedule:
  Serum AMH levels were measured before the stimulation began. Estradiol and FSH levels were measured on the third day of the participants' menstrual cycle. Ovarian stimulation started on the same day with 150 IU of recombinant human Follicle-Stimulating Hormone (r-FSH) after a transvaginal ultrasound was performed, provided that serum FSH levels were below 16 mIU/ml and estradiol levels were under 70 pg/ml (r-FSH group). All patients underwent routine monitoring with transvaginal ultrasound. The GnRH antagonist cetrorelix acetate, at a dose of 0.25 mg/day was given when a dominant follicle reached 14 mm in diameter. Oocyte retrieval (OPU) was performed 34-36 hours after hCG administration followed by IVF/ICSI and embryo transfer on day 3 after OPU
  Interventions: Drug: Clomiphane citrate; Drug: recombinant human Follicle-Stimulating Hormone (r-FSH-alfa)
- High-dose Gonadotropins (r-FSH) (Active Comparator): Patients in this group will be stimulated according to the high-dose short r-FSH antagonist protocol.
  Treatment schedule:
  Ovarian stimulation started on day 3 with 300 IU of recombinant human Follicle-Stimulating Hormone (r-FSH) after a transvaginal ultrasound was performed, provided that serum FSH levels were below 16 mIU/ml and estradiol levels were under 70 pg/ml (r-FSH group). All patients underwent routine monitoring with transvaginal ultrasound and serum estradiol measurements. The GnRH antagonist cetrorelix acetate, at a dose of 0.25 mg/day, was given when a dominant follicle reached 14 mm in diameter. Oocyte retrieval (OPU) was performed 34-36 hours after hCG administration, followed by IVF/ICSI and embryo transfer on day 3 after OPU.
  Interventions: Drug: recombinant human Follicle-Stimulating Hormone (r-FSH-alfa)

INTERVENTIONS:
Drug: Clomiphane citrate — Clomiphene citrate 100mg/day from day 3 to day 7 of the cycle (5 days) will be added to the low-dose (150 IU) short GnRh antagonist protocol (recombinant human Follicle-Stimulating Hormone (r-FSH-alfa) (Gonal-f; Merck Serono Hellas AE))
  Other Names: Clomiphene citrate 50mg/tab; Serpafar 50mg/tab
  Arms: Clomiphene Citrate (CC)/r-FSH
Drug: recombinant human Follicle-Stimulating Hormone (r-FSH-alfa) — All patients will undergo ovarian stimulation with the standard-dose GNRH-antagonist protocol.
  Ovarian stimulation will be initiated with 150 IU of of recombinant human Follicle-Stimulating Hormone (r-FSH-alfa) (Gonal-f; Merck Serono Hellas AE)
  Other Names: Gonal-f 150 Iu/day; Gonal-f 300 IU/day

SUMMARY:
In the present study we examined the effect of addition of CC to a low dose gonadotropin (150 IU/day) / GnRH antagonist protocol in comparison to a high gonadotropin dose (300 IU/day) regiment (short protocol) in women with poor ovarian responce (POR).

DETAILED DESCRIPTION:
22 patients diagnosed with poor ovarian response, aged 35-43 years, were enrolled in the study. The definition of poor response was based on the presence of at least one of the following criteria: Age equal or over 40 years old or other cause of subfertility, AFC less than 5-7, AMH 0.5-1,1ng/ml , a previous POR (≤3 oocytes with a conventional stimulation protocol or cancellation due to poor response) . All patients received appropriate counselling . Early follicular phase FSH and estradiol (E2) were measured prior to the initiation of treatment. All women had measurements of serum FSH and estradiol and a pelvic sonogram on the second day of their cycle. Providing that serum FSH level was less than 16 mIU/ml and estradiol level less than 70 pg/ml on cycle day2 , ovarian stimulation was initiated with 300 IU of gonadotropins either in the form of a combination of highly purified urinary FSH and LH or with a combination of recombinant FSH and recombinant LH. All patients were re-evaluated on day 5 of the stimulation, and dosage adjustments were made and the antagonists (Cetrorelix or ganirelix 0.25 mg/day) were initiated when at least one follicle reached a diameter of 14mm . When at least 2 follicles reached an average diameter of 18 mm, final oocyte maturation was triggered with 10,000IU of hCG ( Ovitrelle, Greece Inc.). Oocyte retrieval was performed 34 to 36 hours later. All patients underwent ICSI. Patients with successful fertilization underwent embryo transfer under sonographic guidance on day 5 after retrieval. Serum β-hCG levels were measured 12 days after oocyte retrieval, and clinical pregnancy was confirmed by transvaginal ultrasound 14 days later. Ongoing pregnancy was confirmed at 12 weeks by ultrasound. In case of negative pregnancy test result the same participants received CC (100 mg/day) from day 3 to day 7 of the menstrual cycle, in combination with low-dose gonadotropins (150 IU/day) until the day of hCG administration. The primary outcome measure was ongoing pregnancy rates. Secondary outcomes included the number of follicles, the number of mature oocytes, fertilization rate, total number of embryos and embryo quality in each group. Furthermore, we included biochemical pregnancy rates and miscarriage as secondary outcomes as well.

ELIGIBILITY:
The inclusion criteria, established by the European Society of Human Reproduction and Embryology (ESHRE), define POR as the presence of at least two of the following features, had to be met:

* Advanced maternal age (≥40 years) or any other risk factor for POR
* A previous POR (≤3 oocytes with a conventional stimulation protocol)
* An abnormal ovarian reserve test (Day 3 follicle-stimulating hormone (FSH) > 12 mIU/ml
* Anti-Müllerian hormone (AMH) < 2ng/ml).

Exclusion Criteria:

The succesful ongoing pregnancy after the first stimulation.

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rates | 28 months from start of study
  succesfull clinical pregnancy after performing ultrasound on 12 weeks of pregnancy

SECONDARY OUTCOMES:
Number of follicles | 24 months from start of study
  Calculated on the day of triggering
Number of mature oocytes | 24 months from start of study
  MII
Fertilization rate | 24 months from start of study
  Percentage
Total number of embryos in each group | 24 months from start of study
  Total number of embryos
Biochemical pregnancy rates | 24 months from start of study
  Absence of clinical pregnancy
Miscarriage rates | 28 months from start of study
  Percentage of pregnancies that did not reach viability

CONTACTS AND LOCATIONS:
Overall Officials: Olga Triantafyllidou, MD,, Principal Investigator — University of Athens School of Medicine
Locations (2):
- Greece (2):
  - Aretaieion University Hospital, Athens, Attica
  - Aretaieion University Hospital, Athens

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pilehvari S, ShahrokhTehraninejad E, Hosseinrashidi B, Keikhah F, Haghollahi F, Aziminekoo E. Comparison Pregnancy Outcomes Between Minimal Stimulation Protocol and Conventional GnRH Antagonist Protocols in Poor Ovarian Responders. J Family Reprod Health. 2016 Mar;10(1):35-42. PMID 27385972
- [Background] Moffat R, Hansali C, Schoetzau A, Ahler A, Gobrecht U, Beutler S, Raggi A, Sartorius G, De Geyter C. Randomised controlled trial on the effect of clomiphene citrate and gonadotropin dose on ovarian response markers and IVF outcomes in poor responders. Hum Reprod. 2021 Mar 18;36(4):987-997. doi: 10.1093/humrep/deaa336. PMID 33367742
- [Background] Liu S, Liu X, Li H, Liu M, Lv Y, Li Y. Clomiphene citrate priming increases sensitivity during ovarian stimulation in poor ovarian responders undergoing in vitro fertilization treatment: a retrospective cohort study. Hum Fertil (Camb). 2023 Dec;26(5):1080-1086. doi: 10.1080/14647273.2022.2109069. Epub 2022 Aug 11. PMID 35950570
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35950570/